CLINICAL TRIAL: NCT06778330
Title: The Effect of Combination of Dapagliflozin and Sildenafil in Treatment of Heart Failure Patients With Secondary Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Abdallah, teaching assistant, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M 722
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure NYHA Class II
MeSH Terms: interventions — dapagliflozin; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Active Comparator)
  Interventions: Drug: Dapagliflozin (DAPA); Drug: Sildenafil
- control group (Active Comparator)
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Control group: receive dapagliflozin in addition to standard therapy
Drug: Sildenafil — Test group: receive combination therapy of dapagliflozin and a small dose of sildenafil(25mg/day) in addition to standard therapy
  Arms: test group

SUMMARY:
This study aims to determine the efficacy of sildenafil (improve PAH) as an add-on therapy to dapagliflozin in the treatment of heart failure patients with secondary pulmonary arterial hypertension and compare the result with monotherapy dapagliflozin

ELIGIBILITY:
Inclusion Criteria:

patients with established heart failure with secondary pulmonary hypertension seen by a primary care provider to diagnose a heart disease, the patient's symptoms which may experience:

* Dizziness or fainting
* Heart palpitations, which may feel like your heart fluttering or skipping beats
* Shortness of breath

Exclusion Criteria:

* Patients with a history of severe allergic reactions or hypersensitivity to sildenafil, dapagliflozin, or related medications.
* Individuals with contraindications to the use of sildenafil or dapagliflozin.
* Patients with pulmonary arterial hypertension (PAH) due to conditions other than heart failure (e.g., idiopathic PAH).
* severe hepatic impairment
* aged less than 18 years.
* valvular heart disease .
* Patients with a known or suspected history of non-compliance with medical treatment or inability to adhere to study procedures.
* life expectancy of less than 6 months .
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
change in ejection fraction | 12 weeks after treatment
  Determine the influence of sildenafil as an add-on to dapagliflozin on Left ventricular ejection fraction using function using echocardiography
change in systolic pulmonary artery pressure | 12 weeks after treatment
  Determine the influence of sildenafil as an add-on to dapagliflozin on systolic pulmonary artery pressure using echocardiography
  * Evaluate the impact of sildenafil as an adjunct therapy to dapagliflozin on pulmonary arterial hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided